CLINICAL TRIAL: NCT00564330
Title: In Vivo Quantification of Dental Demineralisation Using Optical Coherence Tomography Before and After Double-blind, Randomised Treatment With Esomeprazole or Placebo of Patients With Dental Erosions
Brief Title: In Vivo Quantification of Dental Demineralisation Using OCT With and Without Esomeprazole
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brain-Gut Research Group (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: D9612L00118
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Tooth Erosion
Keywords: dental erosion; OCT; proton pump inhibitor
MeSH Terms: conditions — Tooth Erosion | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- esomeprazole (Active Comparator): Esomeprazole 20mg twice daily
  Interventions: Drug: Esomeprazole
- placebo (Placebo Comparator): Placebo tablet twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — 20mg bid
  Other Names: Nexium
  Arms: esomeprazole
Drug: Placebo — Placebo bid
  Arms: placebo

SUMMARY:
Dental erosions in 30 male and female patients with proven abnormal gastrooesophageal reflux will be assessed clinically and using a novel optical coherence tomography (OCT) laser technique before and after double-blind randomization to antisecretory treatment with esomeprazole 20mg or placebo bid for 3 weeks.

The primary objective is to quantify tooth substance loss as well as changes in optical reflectance and scattering of dental hard tissues with and without acid inhibition.

Secondary objectives are:

To compare standardised visual scoring with OCT quantification of reflux damage at the different time points on different teeth.

To assess sex differences in OCT- quantified dental tissue loss.

DETAILED DESCRIPTION:
Dental erosions in 30 male and female patients with proven abnormal gastrooesophageal reflux will be assessed clinically and using a novel optical coherence tomography (OCT) laser technique before and after double-blind randomization to antisecretory treatment with esomeprazole 20mg or placebo bid for 3 weeks.

The primary objective is to quantify tooth substance loss as well as changes in optical reflectance and scattering of dental hard tissues with and without acid inhibition.

Secondary objectives are:

To compare standardised visual scoring with OCT quantification of reflux damage at the different time points on different teeth.

To assess sex differences in OCT- quantified dental tissue loss

ELIGIBILITY:
Inclusion Criteria:

1. Dental erosions with Lussi score greater than 1, diagnosed by dentist
2. Provision of informed consent
3. Male or female aged 18 or above years
4. GORD defined by time with pH<4 greater than 3.5% during 24 hours demonstrated by 24h-hour pH-metry in the last 6 months before the start of the study

Exclusion Criteria:

1. Significant illness within 2 weeks of study begin as judged by investigator.
2. Established or suspected non-reflux causes for dental erosions.
3. Inadequate exclusion of other causes for dental erosions (diet, psychiatric, bruxism, salivary abnormalities, vomiting, etc).
4. Inability or unwillingness to give informed consent.
5. Inability to attend all study.
6. New dental treatment (including dental products) may not be begun from 2 weeks before study begin until the end of the study, except usual dental hygiene with usual toothpaste.
7. Allergy to or other contraindication for treatment with esomeprazole.
8. Use of proton pump inhibitors in 2 weeks or other acid inhibitory drugs in 3 days before study inclusion.
9. Substantial change or planned change in dietary pattern, esp. diets within 2 weeks of study start and for the duration of the entire study.
10. Change or planned change in normal medication or use of herbal, mineral, vitamin preparations within 2 weeks of study start and until the end of the study.
11. Congenital dental defects.
12. Ongoing pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Dental erosions by OCT | 3 weeks

SECONDARY OUTCOMES:
OCT parameters | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clive H. Wilder-Smith, MD, Principal Investigator — Brain-Gut Research Group; Petra Wilder-Smith, Professor, Study Director — Beckman and Laser Institute, University of California, Irvine, USA